CLINICAL TRIAL: NCT05801614
Title: Normalized Glucose Levels in Type 2 Diabetes With Carbohydrate or Caloric Restriction: a Randomized Controlled Trial (CarborCal)
Brief Title: Normalized Glucose Levels in Type 2 Diabetes With Carbohydrate or Caloric Restriction
Acronym: CarborCal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Neda Ekberg, Consultant physician, associate professor, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2020-06848
Record Dates: First submitted 2023-01-02; First posted 2023-04-06 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: Diabetes Mellitus Type 2; Diet; Carbohydrate-Restricted; Caloric restriction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Carb diet (Other): Participants will have acces to a plattform with recepies containing 30 g carbohydrate / day during the first three months and thereafter recepies containing 80 g carbohydrate/ day during the remaining 12 months
  Interventions: Other: Low carb diet
- Low Calori diet (Other): Participants will be asked to by low caloric diet replacement containing 850 kCal/day during the first 3 months, aiming for a weight loss of 10 kg during and thereafter will have access to recepies containing less calorie for weight maintenance during the remaining 12 months
  Interventions: Other: Low carb diet

INTERVENTIONS:
Other: Low carb diet — Low calori diet
  Other Names: Low calori diet

SUMMARY:
This is a randomized controlled trial to determine whether a low-carbohydrate (LC) diet can lead to normalized blood glucose levels in patients with short duration of type 2 diabetes (T2D). Previous studies have shown that caloric restricted diet leading to weight loss can normalize blood glucose levels in approximately 50% of patients with a short duration of diabetes type 2. However, caloric restriction is difficult to maintain. Less restrictive approaches are needed. The hypothesis in this study is that Low carbohydrate diet can results in normalized blood glucose levels in T2D and can be an alternative to caloric restriction diet, both in the shorter term (3 months) and longer term (15 months). The outcome of this study leading to reduction of HbA1c is important for prevention of diabetes complications.

DETAILED DESCRIPTION:
Background Overweight and obesity raise the risk of hyperglycemia which is among the strongest risk factors for morbidity and mortality globally, linked to type 2 diabetes (T2D) as well as, e.g., cardiovascular diseases (CVD), several cancers, dementia, complicated pregnancies and non-alcoholic fatty liver disease.1 The link between obesity, T2D and CVD is partially explained by the visceral adiposity and ectopic (e.g., hepatic) fat associated with insulin resistance, glucose intolerance, arterial stiffness, high blood pressure and dyslipidaemia constituting the metabolic syndrome.2,3 Recent studies have demonstrated that diet-induced weight loss, averaging just over 10 kg at 12-months, can effectively normalize blood glucose levels in T2D in a large proportion of patients. While energy-restrictive diets can enable rapid weight loss, any restrictive diet can be difficult to maintain over time. Strict weight loss diet is difficult to follow. Less restrictive approaches that can be adopted as part of a healthy lifestyle would be ideal.

Cardiovascular complications are the leading cause of morbidity and mortality among patients with diabetes. 29 The mechanisms of diabetes mellitus-associated progression of atherosclerosis are not fully understood. Hyperglycemia has been shown to cause increased oxidative stress arising from oxi-dative degradation of glucose metabolites. Similarly, advanced glycosylation endproducts (AGEs), which are the result of intracellular hyperglycemia, have been shown to be involved in mediating vascular damage. Furthermore hyperglycemia has been reported that to lead to a hypercoagulable state.29 Low carbohydrate diet has recently gained popularity. Rresearch questions remain on if LC diet with low GI can lead to normalization of blood glucose levels and decrease cardiovascular risk markers. The ideal energy percentage (E%) of carbohydrate in the diet for optimal glucose levels is unclear. Caloric restriction diet has shown best results for normalisation of blood glucose levels. There are no previous studies comparing LC diet with caloric restricted diet in regard to normalization of blood glucose levels. The main goal of this study is to evaluate if LC with low GI can lead to normalization or improvement of blood glucose levels in type 2 diabetes (T2D) and to explore the mechanism for normalization of blood glucose levels after LC diet and caloric restricted diet.

The main hypothesis in this study is that Low carbohydrate diet can results in normalization or improvement of blood glucose levels in patients with T2D with short duration of disease both in the shorter term (3 months) and longer term (15 months).

286 patients with type 2 diabetes will be included in this study. Patients will be randomized to a low Carb diet or a low caloric diet for 15 months.

Previous study on caloric restriction diet (DIRECT trial) showed normalization of blood glucose levels in 46% of participants after 12 months. Previous studies on LC diet have shown different results on blood glucose levels based on differences in study design. The greater the carbohydrate restriction, the greater glucose lowering effect. There is a lack of studies reporting normalisation of blood glucose levels. Therefore, it was assumed that LC dietary strategies can result in normalization of blood glucose levels in 30% of patients with T2D after 3 and 15 months. Using an online sample size calculator for a study power of 80% and alpha value of 0.05 the sample size was calculated to 143 participants in each group.

Anthropometric data and blood samples will be collected at baseline and after 3 months (initial weight loss and remission) months (continued weight loss and remission), and 15 months (weight maintenance). For security reason Hb1c and lipid status will be analyzed after changes in medication. For Standardized measurement protocols, instruments (e.g., for anthropometrics), collection tubes, etc. will be used. HbA1c, glucose, lipids and other standard biochemical variables will be measured directly on the day of the visit at the laboratories, or, for substances sensitive to batch effects (e.g., serum insulin), after collection and freezing at -80°C. Samples that are not analyzed immediately will be stored in a biobank for later use. The study will be performed in accordance with GCP.

Controlled diet that leads to weight reduction can reverse type 2 diabetes or delay the diagnosis of T2D. According to the report from the Swedish Institute for Health and Healthcare Economi (IHE) decreasing the blood sugar levels in patient with T2D will spare 800 cases of heart infarction, 500 cases of stroke, 450 cases of kidney failure and 20 cases of blindness. Delaying the diabetes diagnosis is beneficial for the patients since the diabetes complications are directly correlated to the diabetes duration. Patient with type 2 diabetes who change their diet with less carbohydrate have shown to need less insulin. The cost of diabetes disease is affected by the cost of medications and the cost of complications of diabetes. Improved knowledge about which diet can reverse T2D and improve glucose levels will in the end affect the cost for the type 2 diabetes. Dietary intervention which effectively improve blood sugar levels will have significant positive health economic effects. The result from this study will be used for diet recommendation for patients with T2D.

Both men and women will be included in the study. Sex will also be one of the factors in randomisation to assure both groups have equal percent of men and women. Gender is considered a risk factor for obesity. Previous studies have shown that being female doubles the chance of becoming overweight. It is known that lifestyle intervention programs are effective in the prevention of type 2 diabetes mellitus in high-risk populations. However, most studies report poorly about the influence of sex and/or gender effectiveness of these interventions. Male sex is acknowledged as a diabetes risk factor. Men are marginally higher affected by diabetes all over the world. They are diagnosed at younger age and at lower levels of overweight/obesity. Women on the other hand are the majority of participants in weight loss studies (This was also observed this in our study investigating the effect of intermittent fasting). Women show greater weight control involvement and thus seek medical help for weight loss therapy/surgery earlier. It is not known if men and women have different preference for LC-diet or caloric restriction as strategies for weigh maintenance. We will be able to compare the remission rate for T2D in men and women.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 48 mmol/mol (with or without medical treatment);
* less than 6 years since the diagnosis of T2D
* BMI ≥ 27 kg/m2 (≥ 25 kg/m2 for Asians).

Exclusion Criteria:

* Insulin deficiency.
* HbA1c concentration of 12% or more (≥108 mmol/mol),
* treatment with sulphonyl urea or sodium-glucose-cotrasporter2-inhibitor (SGL2-i),
* myocardial infarction within the previous 6 months,
* severe or unstable heart failure
* other severe diseases including cancer, psychiatric/eating disorders, severe depression - substance abuse,
* conditions that may affect the ability of patients to participate in the study

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
non-diabetic HbA1c | After 3 months
  HbA1c below 48 mmol/mol without antidiabetic medication
non diabetic HbA1c | After 15 months
  HbA1c below 48 mmol/mol without antidiabetic medication

SECONDARY OUTCOMES:
Changes in HbA1c | After 3 and 15 months
  Changes in HbA1c from base line to 3 and 15 months
Percent of participants with HbA1c below 48 and 42 mmol/mol | After 3 and 15 months
  Number of participants with HbA1c below 48 and 42 both on and without antidiabetic medication
Changes in Fasting glucose levels | After 3 and 15 months
  Changes in fasting plasma glucose levels after 3 and 15 months
Changes in HOMA-IR | After 3 and 15 months
  Changes in HOMA_IR afte 3 and 15 months
Changes in Insulin secretion | After 3 and 15 months
  Changes in Insulin secretion measured by glucagon stimulation test

CONTACTS AND LOCATIONS:
Overall Officials: Neda Rajamand Ekberg, MD, PhD, Principal Investigator — Region Stockholm
Locations (1):
- Center for diabetes, Academic Specialist center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No